CLINICAL TRIAL: NCT02593942
Title: Effect of Remifentanil Infusion Alone During the Closure Period for Early Emergence and Hemodynamic Stability in Patients Undergoing Supratentorial Craniotomy
Brief Title: Remifentanil Infusion Alone During the Closure Period for Early Emergence Following Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Hatice Ture, Associate Professor, Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YTU-2014
Record Dates: First submitted 2015-10-03; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Supratentorial Neoplasms
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group I (Experimental): remifentanil
  Interventions: Drug: Remifentanil
- group II (Experimental): remifentanil, propofol
  Interventions: Drug: Remifentanil; Drug: Propofol

INTERVENTIONS:
Drug: Remifentanil — 0.1-0.5 mcg/kg/min infusion
  Other Names: Ultiva
Drug: Propofol — 75-200 mcg/kg/min infusion
  Arms: group II

SUMMARY:
Total intravenous anaesthesia using propofol and remifentanil are routinely used drugs for this purpose. The hemodynamic stability and at the same time early emergency are the main goals following neurosurgery. However there is no standard for discontinuation time for manually controlled systems today.

The investigators aimed to study the effect of remifentanil infusion alone for early emergence and hemodynamic stability during the closure period in patients undergoing supratentorial craniotomy.

DETAILED DESCRIPTION:
Adult, American society of Anaesthesiologist score I-II, 80 patients who underwent elective supratentorial craniotomy for tumour resection were randomly assigned to group I or II. In group I; propofol was discontinued during the dural closure. After the propofol was discontinued, remifentanil dose was increased with the guidance of bispectral index spectrum and hemodynamic parameters. In group II; propofol discontinued before the end of the surgery. Time to awakening and extubation time, adverse events, total remifentanil and propofol consumptions and side effects were recorded. Heart rate and blood pressure were recorded during this period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologist physical status I-II
* Glasgow Coma Scale score of 15 points
* Elective supratentorial craniotomy for tumor resection
* Supine position

Exclusion Criteria:

* Obese patient
* Brain tumor greater than 30 mm in diameter
* Postoperative cranial drainage
* Hypertension
* Diabetes mellitus
* Reoperation
* Pregnant
* Breast feeding
* Allergy to the study medications
* History of cranial radiotherapy
* Frontal bone flap
* Intraoperative neuromonitoring

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time of extubation | 3 hours
  After the surgery, starting from three-pin head holder removal, an investigator asked each patient to open his or her eyes, squeeze the investigator's hand. When the patient opened his or her eyes, obeyed commands, resumed adequate respiration, hemodynamically stable and bispectral index spectrum > 70-80 was extubated, and the time will be recorded. The patients will be followed for an expected average of 3 hours.

SECONDARY OUTCOMES:
Heart Rate | 6 hours
  Heart rate per minute was recorded
Mean arterial pressure were recorded | 6 hours
  Mean arterial pressure (mmHg) was recorded
Post-anesthesia awaking time | 3 hours
  Post-anesthesia awaking time assessed as the interval (min:sec)required to

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Ture, MD., Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University Hospital, Istanbul, Turkey (Türkiye)